CLINICAL TRIAL: NCT00304642
Title: A Study to Assess the Pharmacokinetics of Dapivirine (TMC120) Vaginal Microbicide Gel in Healthy HIV-Negative Women.
Brief Title: A Study to Assess the Pharmacokinetics of Dapivirine (TMC120) Vaginal Microbicide Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPM004
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2006-06-02 (Estimated); Status verified 2006-06

CONDITIONS: HIV Infections
Keywords: HIV-1; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Dapivirine; Vaginal Creams, Foams, and Jellies

INTERVENTIONS:
Drug: dapivirine (TMC120) vaginal gel

SUMMARY:
Approximately 18 women will be enrolled in this single-center, double-blind, randomized Phase I study to assess vaginal tissue and fluid levels, plasma levels and pharmacokinetics of dapivirine (TMC120) gel, which will be applied for 10 consecutive days in 18 healthy HIV-negative women ages 18 to 50. Volunteers will be randomized in a 1:1:1 ratio to receive 2.5mL dapivirine vaginal microbicide gel at one of three concentrations.

ELIGIBILITY:
Inclusion Criteria:

* HIV-negative
* Willing to participate and sign and informed consent form.
* Willing to be tested for HIV and to use an experimental vaginal gel.
* Willing to use a reliable form of contraception during the study.
* Willing to undergo pelvic examinations with colposcopy according to the protocol throughout the study.
* Normal cervical assessment.
* Willing to abstain from using any vaginal product (other than the study product).
* Willing to be sexually abstinent from Day 1 until completion of study product use on Day 10.

Exclusion Criteria:

* Currently pregnant or breast-feeding.
* Currently has any clinically detectable abnormality on the vulva, vaginal walls or cervix.
* Currently has laboratory confirmed gonorrhea, chlamydia, trichomonas or syphilis, has Genital Ulcer Disease (GUD) or vaginal candidiasis symptoms; or has an HSV-2 lesion as indicated by clinical diagnosis or laboratory test.
* Symptomatic bacterial vaginosis (BV) and unwilling to undergo treatment.
* Current use of injection drugs.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18
Dates: Start 2005-11

PRIMARY OUTCOMES:
To assess plasma levels and pharmacokinetics of dapivirine applied vaginally. To measure vaginal fluid and vaginal tissue levels of dapivirine at various time after application of the gel.

CONTACTS AND LOCATIONS:
Overall Officials: Zeda Rosenberg, ScD, Study Director — Beijing Immupeutics Medicine Technology Limited
Locations (1):
- Farmovs-Parexel, Bloemfontein, South Africa